CLINICAL TRIAL: NCT05565365
Title: Ultrasound-guided Transversalis Fascia Plane Block Versus Erector Spinae Plane Block for Post-operative Analgesia in Inguinal Hernia Repair Under General Anesthesia: a Randomized Controlled Study
Brief Title: Transversalis Fascia Plane Block Versus Erector Spinae Plane Block for Analgesia in Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Assistant professor of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SM 10 2022
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion; Parapsychology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis fascia plane (TFP) block (Placebo Comparator): Patients will receive unilateral US-TFP block with bupivacaine 15 minutes before skin incision
  Interventions: Procedure: Transversalis fascia plane (TFP) block
- Erector Spinae Plane (ESP) Block (Active Comparator): Patients will receive unilateral US-ESP block with bupivacaine 15 minutes before skin incision
  Interventions: Procedure: Erector Spinae Plane (ESP) Block

INTERVENTIONS:
Procedure: Transversalis fascia plane (TFP) block — Patients will receive unilateral US-TFP block with 0.3 mL/kg bupivacaine 0.25% 15 minutes before skin incision
  Other Names: TFP block
  Arms: Transversalis fascia plane (TFP) block
Procedure: Erector Spinae Plane (ESP) Block — Patients will receive unilateral US-ESP block with 0.3 mL/kg bupivacaine 0.25% 15 minutes before skin incision
  Other Names: ESP Block
  Arms: Erector Spinae Plane (ESP) Block

SUMMARY:
Uncontrolled postoperative pain after inguinal hernia repair increases the incidence of postoperative complications.

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most common surgical procedures in the world. Annually, more than 20 million inguinal hernia repairs are conducted worldwide.

Uncontrolled postoperative pain increases the incidence of postoperative complications. Regional blocks, as a part of multimodal analgesia, can improve pain control in the postoperative period and reduce complications that may arise from using a single mode of analgesia. For example, reliance on opioid analgesia increases the incidence of pruritus, nausea, and vomiting, as well as respiratory depression.

Hebbard first described the ultrasound (US)-guided transversalis fascia plane (TFP) block in 2009. A local anesthetic (LA) injected between the transversus abdominis muscle and its deep investing fascia will block the anterior and the lateral branches of the T12 and L1 nerves.

Erector spinae plane block (ESPB) is a type of facial plane block in which local anesthetic is administered in the plane located between the erector spinae muscle and thoracic transverse process. ESPB blocks the transmission of nociceptive stimuli through the dorsal/ventral rami of the spinal nerve roots, prevents afferent stimuli transmission, and inhibits efferent activation of the sympathetic nervous system and can thus provide both somatic and visceral sensory blockade, which would make it an ideal regional anesthetic technique for abdominal surgery.The effect of ESPB is also achieved through the block of the lateral, posterior, and anterior thoracic wall resulting in multiple levels sensory blocks. Additional proposed mechanism of action could be explained by the epidural spread of the anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Male patients undergoing elective open unilateral inguinal hernia repair under general anesthesia, ASA status I-II, aged from 20 to 65 years old

Exclusion Criteria:

* Contraindications to regional block (coagulopathy, infection at the needle insertion site, or diaphragmatic paralysis)
* Altered cognitive function
* Body mass index (BMI > 35 kg/m2)
* Patients who have difficulty understanding the study protocol
* Patients who have any known allergy to study medications
* Advanced hepatic or renal failure
* Chronic opioid consumption
* Patient refusal

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-14 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
The intensity of postoperative pain | 24 hours after surgery
  Assessed by the verbal analog pain scale graded from 0 to 10 (0 = no pain, and 10 = the worst possible pain)